CLINICAL TRIAL: NCT06308874
Title: A Double-Blind, Placebo Controlled, Single Dosing, Dose-Escalation Phase 1 Clinical Trial to Investigate the Safety, Tolerability, PK/PD of J2H-1702 After Oral Administration in Healthy Female Subjects
Brief Title: Investigate Safety, Tolerability, PK/PD of J2H-1702 in Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: J2H Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JH-222-101
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-02

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Amg dose Group (Experimental): Amg dose administration group
  Interventions: Drug: Amg dose administration group
- Amg dose Group- Placebo (Placebo Comparator): Amg dose administration group- Placebo
  Interventions: Drug: Amg dose administration group- Placebo
- Bmg dose Group (Experimental): Bmg dose administration group
  Interventions: Drug: Bmg dose administration group
- Bmg dose Group- Placebo (Placebo Comparator): Bmg dose administration group- Placebo
  Interventions: Drug: Bmg dose administration group- Placebo

INTERVENTIONS:
Drug: Amg dose administration group — Orally, Amg tablet single administration
  Arms: Amg dose Group
Drug: Amg dose administration group- Placebo — Orally, Placebo Amg tablet single administration
  Arms: Amg dose Group- Placebo
Drug: Bmg dose administration group — Orally, Bmg tablet single administration
  Arms: Bmg dose Group
Drug: Bmg dose administration group- Placebo — Orally, Placebo Bmg tablet single administration
  Arms: Bmg dose Group- Placebo

SUMMARY:
- Objectives: Primary objective_To evaluate the safety and tolerability after single oral administration of the investigational product (IP), J2H-1702 in healthy female subjects. Secondary objective_To evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) characteristics after single oral administration of the IP, J2H-1702 in healthy female subjects.

DETAILED DESCRIPTION:
- Study Methodology: 6 Subjects will be randomized to the study group (J2H-1702 group) and 2 subjects will be to the placebo group. AE, VS, ECG, Lab tests will be evaluated to check the safety, tolerability and PK/PD.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy females aged ≥ 19 and ≤ 45 years
2. Subjects with a body mass index (BMI) ≥ 18.0 to ≤ 27.0 kg/m2
3. Subjects confirmed to be clinically healthy based on the medical history, physical examination, vital signs, electrocardiogram (ECG), and appropriate clinical laboratory tests
4. Agree to use dual contraceptive methods and not to donate eggs
5. Voluntarily agree to participate in the study

Exclusion Criteria:

1. A subject who had or has the disease corresponding to clinically significant liver, etc.
2. A subject with a history of gastrointestinal diseases or surgery
3. A subject who has a history of clinically significant hypersensitivity to drugs containing 11β-HSD1 inhibitor
4. A subject who has genetic problems such as galactose intolerance, Lap galactose intolerance, Lap lactase deficiencies, or glucose ∙galactose malabsorptivity, etc.
5. One who has drug abuse and one who is positive response in urine drug screening tests
6. A subject with abnormal vital signs at the screening visit
7. A subject who has participated in another clinical trial or bioequivalence test
8. A subject who donated whole blood or the ingredient, or received blood transfusion
9. A subject who took drug metabolizing enzyme-inducing and inhibitory drugs
10. A subject who consumes grapefruit/caffeine-containing food
11. A subject who took any prescription drug or herbal medicine or took any Over The Counter Drug (OTC)
12. High caffeine intaker, high alcohol intaker or excessive smoker
13. A subject who cannot eat meals provided by the Clinical Trial institution.
14. A subject who participated in this trial and were administered the investigational product.
15. A subject who is positive for serum test
16. A pregnant or breast-feeding subject
17. A subject who the investigator deems inappropriate for this clinical trial

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Cmax | 1day 0 (Before IP administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours (After IP administration)
  Pharmacokinetics
Emax | -1day 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hours, 1day 0 (Before IP administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24hours (After IP administration)
  Pharmacodynamics

CONTACTS AND LOCATIONS:
Locations (1):
- J2H Biotech, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No